| PROSPECTIVE STUDY INVESTIGATING THE OPTIMAL DURATION OF I | NDWELLING URINARY CATHETER FOLLOWING INFRAPERITONEAL |
|---|---|
| COLORECTAL SURGERY AND ROLE OF | POSTOPERATIVE ALPHA-BLOCKADE |

**Protocol Number:** Version 3 Date 11/30/2012

**Lead Investigator:** Phillip Fleshner, MD

Division of Colorectal Surgery Cedars-Sinai Medical Center

| Protocol No./ Title: | Prospective study investigating the optimal duration of indwelling urinary catheter following infraperitoneal colorectal surgery and role of | |
|---|---|---|
| Statistical Analysis<br>Plan: | postoperative alpha-blockade Determine the incidence of retention of two groups. A control group of 72 hours catheterization (Group 1) to 24 hours catheterization plus medication (Group 2) to potentially reduce retention. | |
| | <b>Data Description</b> : Non-inferiority study p <sub>A</sub> =0.15, p <sub>B</sub> =0.15, d=0.15 (tolerance). We would like to test 1) If Group 2 is non-inferior to Group 1 (2 is not worse than 1). | |
| | Power Analysis and Sample Size Calculation: | |
| | A sample size for 80% power is 71 per group. This would be a total of 142. | |
| | Two group test of equivalence in proportions | |
| | Test significance level, a (one-sided) | 0.050 |
| | Standard proportion, p <sub>S</sub> | 0.150 |
| | Equivalence limit difference,<br>p <sub>T</sub> - p <sub>S</sub> , D <sub>0</sub> | 0.150 |
| | Test expected proportion, p <sub>T</sub> | 0.150 |
| | Expected difference, p <sub>T</sub> - p <sub>S</sub> , D <sub>1</sub> | 0.000 |
| | Power (%) | 80 |
| | n per group | 71 |